CLINICAL TRIAL: NCT00233714
Title: A Randomized Feasibility Study of the Double Dose or Single Dose Sirolimus-Eluting BX VELOCITY Balloon-Expandable Stent for the Treatment of Diabetic Patients With de Novo Native Coronary Artery Lesions(3D)
Brief Title: Double or Single Dose Sirolimus-Eluting Stents in Diabetic Patients With de Novo Coronary Artery Lesions
Acronym: 3D
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sid Cohen, MD, VP, Cordis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P03-6318
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Single-dose Sirolimus-Eluting Coronary stent
  Interventions: Device: CYPHER Sirolimus-Eluting Coronary Stent
- 2 (Active Comparator): Double-dose Sirolimus-Eluting Coronary stent
  Interventions: Device: CYPHER Sirolimus-Eluting Coronary Stent

INTERVENTIONS:
Device: CYPHER Sirolimus-Eluting Coronary Stent — Single dose Sirolimus-Eluting coronary stent
  Other Names: Cypher Bx Velocity
  Arms: 1
Device: CYPHER Sirolimus-Eluting Coronary Stent — Double-dose Sirolimus-Eluting coronary stent
  Other Names: Cypher Bx Velocity
  Arms: 2

SUMMARY:
The main objective of this study is to assess safety and effectiveness of double dose sirolimus-eluting Bx VELOCITY stents in diabetic patients with a de novo native coronary lesion, as compared to single dose sirolimus-eluting Bx VELOCITY™ stents.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be minimum 18 years of age;
2. Patients must be previously diagnosed with diabetes with documented treatment with insulin, oral medications, or diet for a minimum of 3 months;
3. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
4. Treatment of one lesion in a native coronary artery. The treated lesion will be the one with the highest % diameter stenosis by visual estimate. Additional study stents may be used for procedural complications such as dissections. Multivessel treatment is permissible in non-target vessels; however, additional lesions may only be treated with commercial stents. If other non-target lesions are treated with commercial stents during the index procedure, they must be successfully treated prior to the study lesion;
5. The target vessel is 2.5 mm and 3.5mm in diameter (visual estimate);
6. The target lesion is <30 mm in length (visual estimate) located in a native coronary artery;
7. Target lesion stenosis is >50% and <100% (TIMI I) (visual estimate);

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK>2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Patients admitted for treatment of diabetic ketoacidosis > 2 times in the past six months (Brittle Diabetics);
3. Ejection fraction 30%;
4. Impaired renal function (creatinine > 2.0 mg/dL);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-05; Primary Completion 2004-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is in-stent late lumen loss as measured by QCA at 6 months post-procedure. | 6 months post-procedure

SECONDARY OUTCOMES:
Composite of Major Adverse Cardiac Events (MACE) defined as death, myocardial infarction (Q wave and non-Q wave), emergent bypass surgery, or repeat target lesion revascularization at 30 days, 6 months, 12 months and 2, 3, 4 and 5 years post-procedure. | 30 days, 6 months, 12 months and 2, 3, 4 and 5 years post-procedure
Target lesion revascularization (TLR) and target vessel revascularization (TVR) at 30 days, 6 months, 12 months and 2, 3, 4 and 5 years post-procedure. | 30 days, 6 months, 12 months and 2, 3, 4 and 5 years post-procedure
Target vessel failure (TVF) defined as cardiac death, myocardial infarction, or target vessel revascularization at 30 days, 6 months, 12 months and 2, 3, 4 and 5 years post-procedure. | 30 days, 6 months, 12 months and 2, 3, 4 and 5 years post-procedure
Device success defined as achievement of a final residual diameter stenosis of <50% (by QCA), using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used. | During Index Procedure
Lesion success defined as the attainment of <50% residual stenosis (by QCA) using any percutaneous method. | During Index Procedure
Procedure success defined as achievement of a final diameter stenosis of <50% (by QCA) using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay. | During the hospital stay
In-stent and in-lesion binary restenosis (> 50% diameter stenosis) as measured by QCA at 6 months and 2 years. | 6 months and 2 years
In-stent and in-lesion mean percent diameter stenosis (%DS) and minimal lumen. diameter (MLD) measured by QCA post-procedure and at 6 months and 2 years. | post-procedure and at 6 months and 2 years
In-lesion late lumen loss measured by QCA at 6 months and 2 years. | 6 months and 2 years
Stent lumen and stent obstruction volume by intravascular ultrasound (IVUS) at post-procedure and 6 months and 2 years. | post-procedure 6 months and 2 years.
Glycemic control as measured by HbA1c at baseline, 6, 12, and 24 months. | baseline, 6, 12, and 24 months
C-reactive protein levels measured at baseline, 6, 12, and 24 months related to patient outcomes. | baseline, 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose E. Sousa, MD, Principal Investigator — Institute Dante Pazzanese of Cardiology
Locations (1):
- Institute Dante Pazzanese of Cardiology, São Paulo, Brazil

REFERENCES:
- [Result] Costa RA, Sousa JE, Abizaid A, Chaves A, Feres F, Sousa AG, Musumeci G, Mehran R, Fitzgerald PJ, Lansky AJ, Leon MB, Shiran A, Halon DA, Lewis BS, Guagliumi G. The randomised study of the double dose versus single dose sirolimus-eluting stent for the treatment of diabetic patients with de novo coronary lesions. EuroIntervention. 2006 Nov;2(3):295-301. PMID 19755304
- [Result] Hur SH, Ako J, Shimada Y, Tsujino I, Hassan AH, Abizaid A, Shiran A, Lewis BS, Guagliumi G, Cohen SA, Honda Y, Fitzgerald PJ, Sousa JE. Two-year intravascular ultrasound observations in diabetic patients treated with single and double dose sirolimus-eluting stents: results of the double dose diabetes (3D) study. J Invasive Cardiol. 2008 Aug;20(8):411-6. PMID 18688066